CLINICAL TRIAL: NCT04834570
Title: Breast Cancer Survivors: Main Physical and Psychosocial Problems After Completion of Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Thiago Vidal Brito, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Other Study IDs: 32155120.7.0000.0072
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Quality of life; Survivorship; Oncology
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Survivors: Women who have survived breast cancer for at least 1 year (12 months) and 2 years (24 months) after the end of primary treatment
  Interventions: Behavioral: Quality of life in Breast Cancer Survivors

INTERVENTIONS:
Behavioral: Quality of life in Breast Cancer Survivors — The patient will receive the following questionnaires to be completed :
  * EORTC QLQ-C30
  * EORTC QLQ - BR-23
  * FACT-B

SUMMARY:
Breast cancer directly affects women physically, psychologically and socially in the process of diagnosis, treatment and post-treatment. Despite the improvement in conventional breast cancer treatments that led to longer disease-free survival, many patients still suffer from physical, psychological, social and spiritual problems after treatment. The neglect of physical and psychosocial problems faced by patients who are between 1 and 2 years after the end of treatment negatively impacts the quality of life of this population.

DETAILED DESCRIPTION:
The purpose of the study is to assess the overall quality of life and measure the impact on women who have survived breast cancer for at least 1 year (12 months) and 2 years (24 months) after the end of primary treatment and to identify possible repercussions of breast cancer and its treatments associated with Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Adult women (age ≥ 20 years old and less than 60 years old)
* Patient who has been treated by surgery, with or without adjuvant chemotherapy
* Clinical Stages I, II and III
* Patients considered cured, without history of recurrences
* Patients who completed treatment within a minimum of 1 year and are currently being undergoing outpatient follow-up

Exclusion Criteria:

* Initial diagnosis of another type of cancer, other than breast cancer
* Bilateral breast cancer
* Patient unable to fill out the QoL questionnaire
* Patient with disease recurrence
* Patient with metastatic breast cancer

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recruitment of 100 breast cancer patients who have completed treatment within a minimum of 1 year and are currently undergoing outpatient follow-up
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Global Health Status by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire) | 1 year after treatment ends; 2 years after treatment ends;
  This questionnaire was designed to be cancer specific, and includes all emotional, social and physical aspects of the individual's life. The scores in each dimension are uniformly transformed to dimensions ranging from 0 to 100, with 0 denoting the negative (low functioning, high symptom burden) and 100 the positive end (high functioning, low symptom burden) of the continuum.

SECONDARY OUTCOMES:
Quality of life specific for breast cancer by EORTC QLQ-BR23 (European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire) | 1 year after treatment ends; 2 years after treatment ends;
  The questionnaire contains 23-item, two breast cancer specific functional scales (body image and sexuality) and three symptom scales evaluating arm symptoms, breast symptoms, and systemic therapy symptoms. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Quality of life by FACT-B+4 (Functional Assessment of Cancer Therapy-Breast) | 1 year after treatment ends; 2 years after treatment ends;
  The FACT-B+4 questionnaire (Functional Assessment of Cancer Therapy-Breast) consists of 40 questions: 27 about general quality of Life and 13 about breast cancer. It is fur-ther structured into five subscales: physical, family-social, emotional, functional well-being and a last part specific for breast cancer. The result given by the sum of the scores goes from zero to 164: a higher score corresponds to major well-being of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- IBCC Oncologia, São Paulo, Brazil